CLINICAL TRIAL: NCT03457935
Title: The Role of the miR200 Family in the Restoration of Normal Lung Homeostasis and Detection of Early IPF
Brief Title: Detection of Early Idiopathic Pulmonary Fibrosis
Status: Active, not recruiting | Type: Observational
Sponsor: Temple University (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 23201
Record Dates: First submitted 2018-02-28; First posted 2018-03-08 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-09

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Non-IPF ILD: non-IPF ILD diagnosis
  Interventions: Other: blood samples
- IPF: Naive patients with no IPF treatment
  Interventions: Other: blood samples
- Control: no lung diseases
  Interventions: Other: blood samples

INTERVENTIONS:
Other: blood samples — Blood samples

SUMMARY:
The purpose of the study is to determine if miR200 family may serve as a biomarker of IPF.

ELIGIBILITY:
Inclusion Criteria for IPF Patients:

* Informed consent
* Subjects ≥ 40 y.o.
* Naive patients with no IPF treatment
* IPF diagnosis based on the ATS/ERS/JRS/ALAT criteria

Inclusion Criteria for non-IPF ILD Patients:

* Informed consent
* Subjects ≥ 18 y.o.
* ILD diagnosis

Exclusion Criteria:

* HIV
* Hepatitis B
* Hepatitis C
* Pregnant or lactating women

inclusion criteria for controls: informed consent >18 years old; no lung diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with non-IPF ILD and a new diagnosis of IPF.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2018-04-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
To determine miR200 levels (fold change) in blood samples. | Baseline (one time).
  MicroRNAs (miRs) are noncoding small RNAs, which regulate numerous physiological and pathological processes. miR200 levels will be measured in blood samples collected from control subjects, non-IPF ILD and IPF patients. These samples will be used for identifying biomarkers for IPF.

CONTACTS AND LOCATIONS:
Locations (1):
- Temple University, Philadelphia, Pennsylvania, United States